CLINICAL TRIAL: NCT02634866
Title: Multivariate ASSEssment of CardiovascUlar Response to the Controlled Exercise in Patients With Hypertension - Prospective and Observational Study (ASSECURE Study)
Brief Title: Cardiovascular Response to Exercise in Hypertension
Acronym: ASSECURE
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Paweł Krzesiński, Lecturer, Military Institute od Medicine National Research Institute
Other Study IDs: 0000000336
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: hypertension; exercise; diastolic heart failure
MeSH Terms: conditions — Hypertension; Motor Activity; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group N: The subjects with no symptoms of HF and normal left ventricular diastolic function (no less than 40 subjects)
- Group D: The subjects with no symptoms of HF and left ventricular diastolic dysfunction (no less than 40 subjects)
- Group D_HF: The subjects with symptoms of HF and left ventricular diastolic dysfunction (no less than 40 subjects)

SUMMARY:
Arterial hypertension (AH) is an important clinical social and economic problem, related to the increased cardiovascular risk. AH is associated with cardiovascular hemodynamic alterations, including left ventricular diastolic dysfunction (LVddf). In consequence of increased blood pressure, the effectiveness of LV as a blood pump decreases and the symptoms of heart failure (HF) may occur. Thus, the identification of noninvasive markers related with the progression from the asymptomatic AH to LVddf/HFpEF would be beneficial.

Another issue is that the diagnostic difficulties in patients with LVddf and HFpEF stem from the limited possibility to assess the hemodynamic response to exercise. Thus, there is a need for more detailed methods of cardiovascular monitoring while exercise testing.

We hypothesize that some new noninvasive hemodynamic parameters, characterizing left ventricular (LV) function and arterial stiffness, may help to predict the risk of cardiovascular events and future occurrence of LVddf/HFpEF. Moreover, we assume that cardiopulmonary exercise test (CPET), completed with new methods of noninvasive hemodynamic monitoring (impedance cardiography and applanation tonometry), would provide additional value in the assessment of the cardiovascular hemodynamic response to exercise.

The study is intended to verify these hypothesis.

DETAILED DESCRIPTION:
Arterial hypertension (AH) is an important clinical social and economic problem, related to the increased cardiovascular risk.

AH is associated with cardiovascular hemodynamic alterations, including left ventricular diastolic dysfunction (LVddf). In consequence of increased blood pressure, the effectiveness of LV as a blood pump decreases and the symptoms of heart failure (HF), even with preserved ejection fraction (HFpEF), may occur. At the early stage, patients' complaints are not specific and difficult to clinical interpretation. As a consequence, these subjects frequently remain undiagnosed. Thus, the identification of noninvasive markers related with the progression from the asymptomatic AH to LVddf/HFpEF would be beneficial.

Another issue is that the diagnostic difficulties in patients with LVddf and HFpEF stem from the limited possibility to assess the hemodynamic response to exercise. Thus, there is a need for more detailed methods of cardiovascular monitoring while exercise testing.

The investigators hypothesize that some new noninvasive hemodynamic parameters, characterizing left ventricular (LV) function and arterial stiffness, may help to predict the risk of cardiovascular events and future occurrence of LVddf/HFpEF. Moreover, the investigators assume that cardiopulmonary exercise test (CPET), completed with new methods of noninvasive hemodynamic monitoring (impedance cardiography and applanation tonometry), would provide additional value in the assessment of the cardiovascular hemodynamic response to exercise.

Aims:

1. The identification of the new markers of cardiovascular risk in patients with arterial hypertension..
2. The identification of the new markers of progression from normal left ventricular diastolic function to left ventricular diastolic dysfunction.
3. The identification of the new noninvasive markers of progression to symptomatic heart failure.
4. The evaluation of the feasibility and usefulness of new methods of noninvasive hemodynamic monitoring (impedance cardiography and applanation tonometry) in the assessment of the cardiovascular hemodynamic response to exercise.
5. Multivariate assessment of cardiovascular response to the controlled exercise, taking into account left ventricular diastolic function and symptoms of heart failure.
6. The relation between laboratory markers of left ventricular remodeling with resting and exercise (noninvasive) hemodynamics.

The study will be performed in a prospective and observational design. No less than 120 hypertensive subjects will be enrolled.

After recruitment the following assessment will be performed:

* anamnesis and physical examination with anthropometrics (including body composition analysis with use of bioimpedance method);
* electrocardiogram;
* echocardiography (resting), including assessment of left ventricular systolic (2-D left ventricular ejection fraction, longitudinal strain) and diastolic function (including tissue Doppler imaging);
* impedance cardiography (resting);
* Applanation tonometry (resting);
* 24-h Holter-ekg (including heart rate variability analysis);
* 24-h ambulatory blood pressure monitoring;
* flow-mediated dilation of brachial artery (FMD);
* 6-minute walking test (6-MWT);
* Cardiopulmonary exercise test (CPET), supported by hemodynamic monitoring with impedance cardiography and applanation tonometry;
* Quality of life assessment (SF 36 questionnaire);
* Laboratory tests (including creatinine, urea, uric acid, lipids, glucose, microalbuminuria, N-terminal of the prohormone brain natriuretic peptide, galectin-3, copeptin, soluble ST2, Growth differentiation factor 15 (GDF-15), human tissue inhibitor of metalloproteinases 1 (TIMP-1), metalloproteinase 2 (MMP-2), metalloproteinase 9 (MMP-9), syndecan-1).

After 12 months (first control visit) and 24 months (second control visit) the echocardiography and clinical assessment (HF symptoms) will be performed to identify: 1/ patients with new onset LVDdf (among group N); 2/ patients with new onset HF (among group D)

Morover, the follow-up of min 48 months concerning cardiovascular events will be performed (as defined below)

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex
* age 40-75 years
* arterial hypertension diagnosed ≥3 months before recruitment.

Exclusion Criteria:

* office blood pressure > 160/100 mmHg
* coronary artery disease
* systolic heart failure (LVEF below 45%) and/or severe heart defect (i.e. valvular disease)
* severe pulmonary diseases (COPD stage C/D, uncontrolled asthma, pulmonary hypertension, pulmonary embolism)
* chronic kidney disease (MDRD eGFR<60 ml/min/1.73m2)
* severe inflammatory disease
* severe mental and physical disorders
* polyneuropathy
* obesity with BMI > 40 kg/m2
* life expectancy less than 12 months in the opinion of the physician
* patients' refusal to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No less than 120 hypertensive subjects (both sexes, aged 40-75 years) will be enrolled, including those with: 1/ no symptoms of HF and normal LV diastolic function (group N, no less than 40 subjects), 2/ no symptoms of HF and LVddf (group D, no less than 40 subjects), 3/ with symptoms of both HF and LVddf (group D_HF, no less than 40 subjects).
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
complex end-point (death from cardiovascular causes and/or myocardial infarction and/or stroke and/or decompensated heart failure) | 48 months
  Any of the following cardiovascular events: death from cardiovascular causes and/or myocardial infarction and/or stroke and/or decompensated heart failure

SECONDARY OUTCOMES:
death from any cause | 48 months
death from cardiovascular causes | 48 months
myocardial infarction | 48 months
decompensated heart failure | 48 months
stroke | 48 months

OTHER OUTCOMES:
new-onset of heart failure after 12 months (in groups N i D) | 12 months
  based on questionnaire
new-onset of heart failure after 24 months (in groups N i D) | 24 months
  based on questionnaire
new-onset of left ventricular diastolic dysfunction in echocardiography after 12 months (in group N) | 12 months
new-onset of left ventricular diastolic dysfunction in echocardiography after 24 months (in group N) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided